CLINICAL TRIAL: NCT07055763
Title: Effect Of Nigella Sativa Oil for the Treatment of Hypertension
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSAHSW/Batch-Fall23/924
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nigella sativa oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nigella sativa Oil Supplementation (Experimental)
  Interventions: Combination Product: Nigella sativa (black seed)
- No Intervention (Control Group) (No Intervention)

INTERVENTIONS:
Combination Product: Nigella sativa (black seed) — Participants in Group 1 (intervention group) will receive Nigella sativa (black seed) oil at a dosage of 0.5 ml, administered orally twice daily-once before breakfast and once before bedtime-for a duration of 12 weeks. The oil, sourced from a standardized local supplier, is rich in thymoquinone, known for its antioxidant and vasodilatory properties. Blood pressure will be measured at baseline and biweekly intervals using a calibrated digital sphygmomanometer to monitor changes in systolic and diastolic values. Participants will also be monitored regularly for any adverse effects.
  Arms: Nigella sativa Oil Supplementation

SUMMARY:
My research explores the antihypertensive effects of Nigella sativa (black seed) oil in managing high blood pressure. Hypertension is a growing global health concern, often insufficiently controlled by standard medications. Nigella sativa, known for its bioactive compound thymoquinone, possesses antioxidant, anti-inflammatory, and vasodilatory properties, making it a potential natural remedy for blood pressure regulation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 to 70 years
* Diagnosed with mild to moderate hypertension (BP ≥140/90 mmHg)
* Willing to participate and provide written informed consent
* Not currently on any herbal or nutritional supplements

Exclusion Criteria:

* History of smoking or alcohol consumption
* Pregnant, postmenopausal, or breastfeeding women
* Use of dietary supplements or medications containing antioxidants, caffeine, estrogen, or steroids
* Individuals engaging in regular vigorous physical exercise
* Those adding extra salt to their meals
* Known allergy to Nigella sativa or black seed oil

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Structured Patient History Questionnaire | 12 Months
  A pre-designed, structured questionnaire will be used at baseline to collect demographic information, medical history, medication use, dietary habits, and lifestyle factors. This is a qualitative tool without a scoring system but is essential for eligibility confirmation and contextual analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria Town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No